CLINICAL TRIAL: NCT02918149
Title: A Randomized Controlled Trial of Ultrasound-Assisted Versus Traditional Landmark Lumbar Puncture in the Neonatal and Infant Population
Brief Title: Ultrasound Assisted Lumbar Puncture in the Neonate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-012757
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Lumbar Puncture
Keywords: Ultrasonography; Infant; Newborn; Lumbar puncture; Spinal puncture; Cerebrospinal fluid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palpation Landmark Technique LP (Other): Traditional landmark palpation technique will be used to perform LP
  Interventions: Other: Palpation Landmark Technique
- Ultrasound-Assisted Technique LP (Experimental): Bedside ultrasonography exam will be used for identification of anatomic landmarks before performing LP
  Interventions: Device: Ultrasound-Assisted Technique LP

INTERVENTIONS:
Other: Palpation Landmark Technique — Clinician will follow routine palpation landmark technique procedure for LP, such as identification of anatomic landmarks by palpation (i.e., superior borders of the posterior iliac crest lies in parallel with L4 spinous process). Palpation will be followed by "blind" stick of the appropriate inter-spinous process space. The study member will have 2 attempts to complete the LP. A "successful" attempt is obtaining cerebrospinal fluid.
  Other Names: Non-Ultrasound Assisted LP
  Arms: Palpation Landmark Technique LP
Device: Ultrasound-Assisted Technique LP — Clinician will use an ultrasound-assisted technique to perform the LP. The Phillips CX50 ultrasound machine is an FDA approved device and will be used in accordance with its approved labeling. Spinal ultrasound will be performed using a linear high-frequency transducer to locate and mark the termination of the conus medullaris, the narrowing of the spinal canal, and the midline to delineate a "safe zone". The study team member will have 2 attempts to complete the LP. A "successful" attempt is obtaining cerebrospinal fluid.
  Other Names: Phillips CX50
  Arms: Ultrasound-Assisted Technique LP

SUMMARY:
Clinicians are often unable to successfully do a spinal tap. Ultrasound has been proposed as a method to improve success but it is not known if it helps. This study is designed to see if ultrasound improves the success rate.

DETAILED DESCRIPTION:
Obtaining cerebrospinal fluid (CSF) through a lumbar puncture (LP) is an essential procedure in the neonatal/infant intensive care unit (N/IICU) for establishing diagnosis and determining treatment. The traditional technique for performing an LP involves palpation of anatomic landmarks followed by a "blind" stick of the appropriate inter-spinous process space. This technique has a failure rate (defined as the inability to obtain cerebrospinal fluid or obtaining a traumatic puncture) of 15-50%.

Bedside ultrasonography possesses the ability to visualize the anatomic landmarks, including the subarachnoid space. In the adult literature, ultrasound has been shown to reduce the LP failure rate. Its utility has also been shown to significantly improve success rates and accuracy in epidural needle placement in neonates and children undergoing regional anesthesia. Increasing the proportion of successful LPs in the N/IICU could significantly reduce patient/family discomfort, sedation exposure, off unit travel, additional interventional procedures and antibiotic use. However, research on the utility of bedside ultrasound assisted LPs by clinicians working in an N/IICU is lacking.

This is a prospective randomized controlled trial. Eligible subjects will be randomized to undergo LP (performed as part of their standard of care) with ultrasound assisted method or traditional landmark method.

Primary Objective:

-To determine if bedside ultrasound-assisted LP, performed by N/IICU clinicians on neonates and infants aged ≤6 months, increases the proportion of successful first attempt non-traumatic LPs when compared to a traditional landmark palpation technique.

Secondary Objectives:

* To determine if bedside-ultrasound assisted LPs increases the proportion of overall successful non-traumatic LPs within 2 attempts.
* To determine if bedside-ultrasound assisted LPs is associated with a decrease in the length of antibiotic exposure in patients undergoing LPs.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates and infants aged ≤6 months
2. Clinical indication for a lumbar puncture (LP), as determined by the clinical team
3. Availability of study personnel to perform bedside ultrasound

Exclusion Criteria:

1. Known spinal cord abnormality (for e.g., tethered cord, spina bifida)
2. Presence of skin and soft tissue infection at insertion site
3. Recent failed LP traumatic LP attempts within the preceding 48 hours
4. Recent diagnosis of intraventricular hemorrhage, within the preceding 7 days
5. Clinically unstable patient, as determined by the clinical team
6. Eligible patients on the resident care team

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Estimated)
Dates: Start 2016-09; Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of successful first attempt LPs | Up to 30 minutes
  The proportion of successful first attempt LPs (defined as obtainment of CSF and non-traumatic LP) for patients in the ultrasound-assisted group compared to the traditional landmark palpation group.

SECONDARY OUTCOMES:
Proportion of overall success of LPs within 2 attempts | Up to 30 minutes
  The proportion of successful first attempt LPs (defined as obtainment of CSF and non-traumatic LP) for patients in the ultrasound-assisted group compared to the traditional landmark palpation group. Providers will have 2 attempts to complete the LP. If CSF cannot be obtained within 2 attempts, any subsequent attempt will be at the discretion of the attending neonatologist and will be performed outside this study by the care team.
Difference in length of antibiotic exposure | Length of Hospitalization (approximately 1 month)
  To determine whether bedside-ultrasound assisted LPs are associated with a decrease in the length of antibiotic exposure in patients undergoing LPs. If LP is unsuccessful, the mean length of antibiotic exposure as compared to patients with successful LPs will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Stoller, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No